CLINICAL TRIAL: NCT04188379
Title: A Phase 3, Multicenter, Randomized, Double-Blinded, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Efgartigimod (ARGX 113) 10 mg/kg Intravenous in Adult Patients With Primary Immune Thrombocytopenia
Brief Title: A Study to Assess the Efficacy and Safety of Efgartigimod in Adult Patients With Primary Immune Thrombocytopenia (ITP).
Acronym: ADVANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-1801; 2019-002100-41 (EudraCT Number)
Record Dates: First submitted 2019-12-04; First posted 2019-12-05 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: immune thrombocytopenia; sustained platelet count response; bleeding events
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — efgartigimod alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- efgartigimod (Experimental): Patient receiving efgartigimod
  Interventions: Biological: efgartigimod
- Placebo (Placebo Comparator): Patients receiving placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: efgartigimod — Intravenous infusion of efgartigimod
  Other Names: ARGX-113
  Arms: efgartigimod
Other: Placebo — Intravenous infusion of placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind placebo-controlled multicenter phase 3 trial to evaluate the efficacy and safety of ARGX-113 in participants with primary ITP.

ELIGIBILITY:
Inclusion criteria:

* Ability to understand the requirements of the trial, to provide written informed consent (including consent for the use and disclosure of research-related health information), and to comply with the trial protocol procedures (including required trial visits).
* Male or female patient aged ≥18 years.
* Confirmed ITP diagnosis, at least 3 months before randomization and according to the American Society of Hematology Criteria, and no known other etiology for thrombocytopenia.
* Diagnosis supported by a response to a prior ITP therapy (other than thrombopoietin receptor agonists [TPO-RAs]), in the opinion of the investigator.
* Mean platelet count of <30×10E9/L from 2 counts: 1 platelet count collected during the screening period and the predose platelet count on the day of randomization.
* At the start of the trial, the patient is either on concurrent ITP treatment(s) and has received at least 1 prior therapy for ITP in the past, or the patient is not on treatment for ITP but has received at least 2 prior treatments for ITP. Patients receiving permitted concurrent ITP treatment(s) at baseline, must have been stable in dose and frequency for at least 4 weeks prior to randomization.
* Women of childbearing potential must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at baseline before trial medication (infusion) can be administered.
* Women of childbearing potential should use a highly effective or acceptable method of contraception during the trial and for 90 days after the last administration of the IMP.

Exclusion criteria:

* ITP/thrombocytopenia associated with another condition, eg, lymphoma, chronic lymphocytic leukemia, viral infection, hepatitis, induced or alloimmune thrombocytopenia, or thrombocytopenia associated with myeloid dysplasia.
* Use of certain medications before the start of the studies (more details in the protocol)
* Patients who have a history of malignancy, including malignant thymoma, or myeloproliferative or lymphoproliferative disorders, unless deemed cured by adequate treatment with no evidence of recurrence for ≥3 years before screening. Patients with completely excised non-melanoma skin cancer (such as basal cell carcinoma or squamous cell carcinoma) or cervical carcinoma in situ would be permitted at any time.
* Uncontrolled hypertension, defined as a repeated elevated blood pressure exceeding 160 mmHg (systolic) and/or 100 mmHg (diastolic) despite appropriate treatments.
* History of any major thrombotic or embolic event within 12 months prior to randomization.
* History of coagulopathy or hereditary thrombocytopenia or a family history of thrombocytopenia.
* History of a recent or planned major surgery (that involves major organs eg, brain, heart, lung, liver, bladder, or gastrointestinal tract) within 4 weeks of randomization.
* Positive serum test at screening for an active viral infection with any of the following conditions: Hepatitis B virus (HBV), Hepatitis C virus (HCV), Human immunodeficiency virus (HIV)
* Clinical evidence of significant unstable or uncontrolled acute or chronic diseases other than ITPdespite appropriate treatments which could put the patient at undue risk.
* Patients with known medical history of hypersensitivity to any of the ingredients of the IMP.
* Patients who previously participated in a clinical trial with efgartigimod and have received at least 1 administration of the IMP.
* Pregnant or lactating females. More details in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (121):
- United States (9):
  - Investigator Site 0010038, Tucson, Arizona
  - Investigator Site 0010045, Washington D.C., District of Columbia
  - Investigator Site 0010034, Jacksonville, Florida
  - Investigator site 0010037, Ocala, Florida
  - Investigator Site 0010042, Iowa City, Iowa
  - Investigator Site 0010046, Greenville, North Carolina
  - Investigator Site 0010049, Cleveland, Ohio
  - Investigator Site 0010040, Columbus, Ohio
  - Investigator Site 0010041, Philadelphia, Pennsylvania
- Austria (3):
  - Investigator Site 0430004, Linz
  - Investigator Site 0430002, Vienna
  - Investigator Site 0430003, Vienna
- Belgium (6):
  - Investigator Site 0320012, Brasschaat
  - Investigator Site 0320011, Bruges
  - Investigator Site 0320015, Leuven
  - Investigator Site 0320014, Turnhout
  - Investigator Site 0320020, Verviers
  - Investigator site 0320002, Yvoir
- Bulgaria (2):
  - Investigator Site 3590001, Pleven
  - Investigator Site 3590002, Sofia
- Czechia (4):
  - Investigator Site 4200001, Brno
  - Investigator Site 4200008, Olomouc
  - Investigator Site 4200006, Ostrava
  - Investigator Site 4200007, Prague
- France (7):
  - Investigator Site 0330019, Clermont-Ferrand
  - Investigator Site 0330009, Créteil
  - Investigator Site 0330015, Le Mans
  - Investigator Site 0330018, Montpellier
  - Investigator Site 0330008, Pessac
  - Investigator Site 0330016, Périgueux
  - Investigator Site 0330017, Rouen
- Georgia (6):
  - Investigator Site 9950006, Tbilisi
  - Investigator Site 9950007, Tbilisi
  - Investigator Site 9950008, Tbilisi
  - Investigator Site 9950009, Tbilisi
  - Investigator Site 9950011, Tbilisi
  - Investigator Site 9950012, Tbilisi
- Germany (3):
  - Investigator Site 0490010, Düsseldorf
  - Investigator Site 0490008, Essen
  - Investigator Site 0490012, Giessen
- Hungary (5):
  - Investigator Site 0360004, Budapest
  - Investigator Site 0360006, Debrecen
  - Investigator Site 0360015, Győr
  - Investigator site 0360010, Nyíregyháza
  - Investigator Site 0360014, Szombathely
- Italy (12):
  - Investigator Site 0390012, Campobasso
  - Investigator Site 0390014, Milan
  - Investigator Site 0390020, Monza
  - Investigator Site 0390015, Novara
  - Investigator Site 0390010, Ravenna
  - Investigator Site 0390011, Reggio Calabria
  - Investigator Site 0390018, Reggio Emilia
  - Investigator Site 0390019, Rimini
  - Investigator Site 0390021, Roma
  - Investigator Site 0390009, Siena
  - Investigator Site 0390017, Torino
  - Investigator Site 0390016, Trieste
- Japan (13):
  - Investigator Site 0810024, Bunkyō City
  - Investigator Site 0810015, Hirakata
  - Investigator Site 0810010, Hiroshima
  - Investigator site 0810017, Iruma
  - Investigator site 0810011, Isehara
  - Investigator Site 0810022, Kashiwa
  - Investigator site 0810018, Maebashi
  - Investigator site 0810020, Minatoku
  - Investigator Site 0810021, Niigata
  - Investigator site 0810014, Sapporo
  - Investigator site 0810016, Shibukawa
  - Investigator Site 0810023, Shimotsuke
  - Investigator Site 0810025, Shinjuku-Ku
- Netherlands (3):
  - Investigator Site 0310005, Rotterdam
  - Investigator Site 0310007, Rotterdam
  - Investigator site 0310006, The Hague
- Poland (10):
  - Investigator Site 0480030, Bialystok
  - Investigator Site 0480015, Brzozów
  - Investigator Site 0480010, Bydgoszcz
  - Investigator Site 0480013, Chorzów
  - Investigator Site 0480012, Gdansk
  - Investigator Site 0480008, Katowice
  - Investigator Site 0480011, Lodz
  - Investigator Site 0480014, Lublin
  - Investigator site 0480026, Nowy Sącz
  - Investigator Site 0480016, Wroclaw
- Russia (6):
  - Investigator site 0070006, Kaluga
  - Investigator Site 0070007, Petrozavodsk
  - Investigator Site 0070013, Rostov-on-Don
  - Investigator Site 0070015, Syktyvkar
  - Investigator Site 0070012, Tula
  - Investigator site 0070010, Ufa
- Spain (10):
  - Investigator Site 0340006, Barcelona
  - Investigator Site 0340007, Barcelona
  - Investigator Site 0340030, Burgos
  - Investigator Site 0340009, Madrid
  - Investigator Site 0340014, Madrid
  - Investigator Site 0340015, Madrid
  - Investigator site 0340012, Palma de Mallorca
  - Investigator Site 0340013, Seville
  - Investigator Site 0340004, Valencia
  - Investigator Site 0340011, Valencia
- Turkey (Türkiye) (16):
  - Investigator Site 0900002, Adana
  - Investigator Site 0900007, Adapazarı
  - Investigator Site 0900003, Ankara
  - Investigator Site 0900006, Ankara
  - Investigator Site 0900008, Ankara
  - Investigator Site 0900015, Ankara
  - Investigator Site 0900016, Edirne
  - Investigator Site 0900013, Istanbul
  - Investigator Site 0900004, Izmir
  - Investigator Site 0900014, Kocaeli
  - Investigator Site 0900018, Malatya
  - Investigator Site 0900005, Manisa
  - Investigator Site 0900010, Mersin
  - Investigator Site 0900009, Samsun
  - Investigator Site 0900017, Tekirdağ
  - Investigator Site 0900019, Trabzon
- Ukraine (2):
  - Investigator Site 3800022, Kharkiv
  - Investigator site 3800006, Mykolayiv
- United Kingdom (4):
  - Investigator Site 0440008, London
  - Investigator Site 0440010, Rhyl
  - Investigator Site 0440012, Southampton
  - Investigator Site 0440014, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Broome CM, McDonald V, Miyakawa Y, Carpenedo M, Kuter DJ, Al-Samkari H, Bussel JB, Godar M, Ayguasanosa J, De Beuf K, Rodeghiero F, Michel M, Newland A; ADVANCE Investigator Study Group. Efficacy and safety of the neonatal Fc receptor inhibitor efgartigimod in adults with primary immune thrombocytopenia (ADVANCE IV): a multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2023 Nov 4;402(10413):1648-1659. doi: 10.1016/S0140-6736(23)01460-5. Epub 2023 Sep 28. PMID 37778358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 71 active sites that enrolled participants in 18 countries. Recruitment started on 09 December 2019.
Pre-assignment Details: During the screening period (up to 2 weeks) the participant's eligibility for trial participation was evaluated. A total of 205 participants were screened, of which 74 participants were screen failures. 131 of 205 were enrolled and randomized at a ratio of 2:1 to receive efgartigimod or placebo.
Groups:
- Efgartigimod: Participants receiving efgartigimod
  efgartigimod: The participants entered a 24-week treatment period and were randomized to receive efgartigimod 10mg/kg IV , weekly from visits 1 to 4 and then from visits 5 to 16 either weekly or q2w, adjusted according to their platelet counts. From visits 17 to 24, subjects were fixed on the dosing schedule at visit 16 or at the last visit at which IMP was administered (ie, either weekly or q2w).
- Placebo: Participants receiving placebo
  Placebo: The participants entered a 24-week treatment period and were randomized to receive placebo IV, weekly from visits 1 to 4 and then from visits 5 to 16 either weekly or q2w, adjusted according to their platelet counts. From visits 17 to 24, participants were fixed on the dosing schedule at visit 16 or at the last visit at which IMP was administered (ie, either weekly or q2w).
Period: Overall Study
Arm/Group | Efgartigimod | Placebo
Started | 86 | 45
Completed | 64 | 32
Not Completed | 22 | 13
Not completed — Withdrawal by Subject | 10 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 3 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Lack of Efficacy | 8 | 5
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All randomized participants.
Groups:
- Efgartigimod: Participants receiving efgartigimod
  efgartigimod: The participants entered a 24-week treatment period and were randomised to receive efgartigimod 10mg/kg intravenous (IV). The investigational medicinal product (IMP) infusion (efgartigimod) was administered weekly from visits 1 to 4, either weekly or every other week (q2w) from visits 5 to 16, and fixed on the dosing schedule of visit 16 (or the last visit at which IMP was administered) from visits 17 to 24 (ie, either weekly or q2w).
- Placebo: Participants receiving placebo
  Placebo: The participants entered a 24-week treatment period and were randomized to receive placebo intravenous (IV). The placebo infusion was administered weekly from visits 1 to 4, either weekly or q2w from visits 5 to 16, and fixed on the dosing schedule of visit 16 (or the last visit at which placebo was administered) from visits 17 to 24 (ie, either weekly or q2w).
- Total: Total of all reporting groups
Arm/Group | Efgartigimod | Placebo | Total
Number analyzed (Participants) | 86 | 45 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 32 | 107
  >=65 years | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (16.55) | 51.7 (17.93) | 48.6 (17.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 24 | 71
  Male | 39 | 21 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 80 | 41 | 121
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 77 | 40 | 117
  Japanese | 5 | 3 | 8
  Unknown or Not reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Chronic ITP With a Sustained Platelet Count Response Defined as Achieving Platelet Counts of at Least 50×10^9/L for at Least 4 of the 6 Visits Between Week 19 and 24 of the Trial.
Description: Percentage of participants with chronic ITP with a sustained platelet count response was defined as achieving platelet counts of at least 50 × 10^9/L for at least 4 of the 6 visits between Week 19 and 24 of the study.
Time Frame: From Week 19 up to Week 24
Population: Full Analysis Set-Chronic population: all randomized participants with chronic ITP.
Measure: Number; unit: Percentage of participants
Groups:
- Efgartigimod: Participants receiving efgartigimod
  Efgartigimod: The participants entered a 24-week treatment period and were randomized to receive efgartigimod 10mg/kg IV, weekly from visits 1 to 4 and then from visits 5 to 16 either weekly or q2w, adjusted according to their platelet counts. From visits 17 to 24, subjects were fixed on the dosing schedule at visit 16 or at the last visit at which IMP was administered (ie, either weekly or q2w).
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 78 | 40
Percentage of participants | 21.8 | 5.0
Statistical Analysis 1: Comparison: Efgartigimod vs Placebo; Test type: Superiority; p = 0.0316, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.884, 95% CI 2-sided [1.007 to 43.591]

2. Secondary Outcome: Extent of Disease Control Defined as the Number of Cumulative Weeks Over the Planned 24-week Treatment Period With Platelet Counts of ≥50×10^9/L in the Chronic ITP Population
Description: Extent of disease control, defined as the cumulative number of weeks over the planned 24-week treatment period with platelet counts of ≥50 × 10^9/L in the chronic ITP population.
Time Frame: From Week 1 up to Week 24
Population: Full Analysis Set-Chronic population: all randomized participants with chronic ITP.
Measure: Median (Inter-Quartile Range); unit: Weeks
Groups:
- Efgartigimod: Participants receiving efgartigimod
  Efgartigimod: The participants entered a 24-week treatment period and were randomized to receive efgartigimod 10mg/kg IV, weekly from visits 1 to 4 and then from visits 5 to 16 either weekly or q2w, adjusted according to their platelet counts. From visits 17 to 24, participants were fixed on the dosing schedule at visit 16 or at the last visit at which IMP was administered (ie, either weekly or q2w).
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 78 | 40
Weeks | 2.00 [0.00 to 11.00] | 0.00 [0.00 to 1.00]
Statistical Analysis 1: Comparison: Efgartigimod vs Placebo; Test type: Superiority; p = 0.0009, Wilcoxon (Mann-Whitney); Median Difference (Net) = 1.000, 95% CI 2-sided [0.000 to 4.000]

3. Secondary Outcome: Percentage of Participants With a Sustained Platelet Count Response for at Least 4 of the 6 Visits Between Week 19 and 24 of the Study
Description: Percentage of participants in the overall population (chronic and persistent ITP) with a sustained platelet count response, defined as achieving platelet counts of at least 50 × 10^9/L for at least 4 of the 6 visits between weeks 19 and 24 of the study.
Time Frame: From Week 19 up to Week 24
Population: Full Analysis Set: all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 86 | 45
Percentage of participants | 25.6 | 6.7
Statistical Analysis 1: Comparison: Efgartigimod vs Placebo; Test type: Superiority; p = 0.0108, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.224, 95% CI 2-sided [1.268 to 26.268]

4. Secondary Outcome: Incidence and Severity of the WHO-classified Bleeding Events
Description: Incidence of the World Health Organization (WHO)-classified bleeding events in the overall population.
  This secondary endpoint used the WHO-classified bleeding scale. Bleeding was the predominant clinical manifestation of ITP and was typically related to platelet count. Accordingly, measuring bleeding was important for monitoring this participant population.
Time Frame: From Week 1 to Week 24
Population: Full Analysis Set: all randomized participants.
Measure: Median (Inter-Quartile Range); unit: bleeding events
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 86 | 45
bleeding events | 4.0 [1.0 to 10.0] | 5.0 [2.0 to 14.0]
Statistical Analysis 1: Comparison: Efgartigimod vs Placebo; Test type: Superiority; p = 0.8287, Wald Test; Rate Ratio = 0.958, 95% CI 2-sided [0.651 to 1.41]

5. Secondary Outcome: Percentage of Participants in the Overall Population Achieving Platelet Counts of at Least 50×10^9/L for at Least 6 of the 8 Visits Between Week 17 and Week 24
Description: Percentage of participants in the overall population achieving platelet counts of at least 50 × 10^9/L for at least 6 of the 8 visits between Week 17 and 24 of the study.
Time Frame: From Week 17 up to Week 24
Population: Full Analysis Set: all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 86 | 45
Percentage of participants | 22.1 | 6.7
Statistical Analysis 1: Comparison: Efgartigimod vs Placebo; Test type: Superiority; p = 0.0265, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.354, 95% CI 2-sided [1.0480 to 22.865]

ADVERSE EVENTS:
Time Frame: Full study duration (31 Weeks).
Description: Treatment emergent adverse events are defined as adverse events starting on or after first administration of any study drug. Safety analyses were performed on the safety analysis set which included all participants in the randomized population who received at least 1 dose or part of a dose of IMP.
Arm/Group | Efgartigimod | Placebo
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/45
Serious Adverse Events (participants affected / at risk) | 7/86 | 7/45
Other Adverse Events (participants affected / at risk) | 80/86 | 43/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efgartigimod (N=86) | Placebo (N=45)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efgartigimod (N=86) | Placebo (N=45)
Haematoma (Vascular disorders) | 8 (17) | 11 (34)
Hypertension (Vascular disorders) | 5 (6) | 0 (0)
Asthenia (General disorders) | 6 (8) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 5 (9) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (24) | 8 (12)
Blood urine present (Investigations) | 31 (66) | 17 (32)
Contusion (Injury, poisoning and procedural complications) | 17 (52) | 6 (42)
Headache (Nervous system disorders) | 14 (20) | 6 (22)
Anaemia (Blood and lymphatic system disorders) | 6 (8) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 2 (7) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 4 (6)
Gingival bleeding (Gastrointestinal disorders) | 4 (6) | 6 (12)
Mouth haemorrhage (Gastrointestinal disorders) | 7 (13) | 7 (10)
Oral blood blister (Gastrointestinal disorders) | 2 (3) | 3 (7)
Nausea (Gastrointestinal disorders) | 5 (9) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 5 (10) | 6 (13)
Petechiae (Skin and subcutaneous tissue disorders) | 13 (21) | 12 (20)
Purpura (Skin and subcutaneous tissue disorders) | 7 (12) | 4 (12)
Haematuria (Renal and urinary disorders) | 14 (30) | 6 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
COVID-19 (Infections and infestations) | 7 (7) | 2 (2)

LIMITATIONS AND CAVEATS:
No limitations reported for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT04188379/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT04188379/SAP_001.pdf